CLINICAL TRIAL: NCT06842303
Title: Contribution of New Pancreatic MRI Sequences for the Evaluation of Tumor Response in Pancreatic Adenocarcinomas
Acronym: PADME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LECLERC Julie, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A01375-42
Record Dates: First submitted 2025-02-03; First posted 2025-02-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pancreas Adenocarcinomas
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patient with a resectable pancreatic lesion (Experimental): Pancreatic resection surgery
  Interventions: Device: Magnetic resonance elastography (MRE).; Device: High-resolution diffusion sequence in MRI
- Patient with a borderline pancreatic lesion (Experimental): Potential pancreatic resection surgery after chemotherapy.
  Interventions: Device: Magnetic resonance elastography (MRE).; Device: High-resolution diffusion sequence in MRI
- Patient with locally advanced pancreatic lesion. (Experimental): Chemotherapy treatment.
  Interventions: Device: Magnetic resonance elastography (MRE).; Device: High-resolution diffusion sequence in MRI

INTERVENTIONS:
Device: Magnetic resonance elastography (MRE). — Magnetic resonance elastography (MRE) is an imaging technique that measures tissue stiffness by assessing the deformation waves produced under external pressure
Device: High-resolution diffusion sequence in MRI — High-resolution diffusion sequence in MRI is an imaging technique that uses the movement of water molecules within tissues to generate detailed images.

SUMMARY:
Pancreatic adenocarcinoma is the most pessimistic digestive cancer in terms of prognosis. Tumor response assessment is crucial, and the recent development of new magnetic resonance imaging sequences, such as high resolution applied to diffusion sequences (Harder et al., 2022) or magnetic resonance elastography (MRE) (Steinkohl et al., 2021), could help address this issue.

ELIGIBILITY:
Inclusion Criteria:

* CT scan diagnosis of non-metastatic pancreatic cancer on contrast-enhanced thoraco-abdomino-pelvic CT;
* Adult patient: age ≥ 18 years;
* Patient affiliated with a social security system or beneficiary of such a system;
* Patient who has received complete information about the research organization and has signed an informed consent form.

Exclusion Criteria:

* Patient with a contraindication to MRI.
* Person referred to in Articles L. 1121-5, L. 1121-7, and L. 1121-8 of the French Public Health Code.

  * Pregnant woman, parturient, or breastfeeding mother;
  * Minor (non-emancipated) individual;
  * Adult individual under legal protection (guardianship, curatorship, or judicial safeguard);
  * Adult individual unable to express consent.
* Person deprived of liberty by a judicial or administrative decision, or person undergoing psychiatric care pursuant to Articles L. 32-12-1 and L. 3213-1 of the French Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2027-06-06 (Estimated)

PRIMARY OUTCOMES:
Absolute elasticity value of the tumor (kPa) before treatment. | Baseline (J0) before treatment
  The absolute elasticity value of the tumor corresponds to the average elasticity value measured within the region of interest, which will be outlined according to the tumor's boundaries.
Absolute elasticity value of the tumor (kPa) after chemotherapy. | 3 months, after chimiotherapy
  The absolute elasticity value of the tumor corresponds to the average elasticity value measured within the region of interest, which will be outlined according to the tumor's boundaries.

SECONDARY OUTCOMES:
For patient with a resectable pancreatic lesion, evaluation of the association between size of the tumor (mm) with the absolute elasticity value of the tumor (kPa). | 3 months, after surgery
For the patients who underwent surgery, evaluation of the association between size of the tumor (mm) and the absolute elasticity value of the tumor (kPa) before chimiotherapy. | 6 months, after surgery
For the patients who underwent surgery, evaluation of the association between size of the tumor (mm) and the absolute elasticity value of the tumor (kPa) after chimiotherapy.. | 6 months, after surgery
For patient with a resectable pancreatic lesion, evaluation of the association between size of the tumor (mm) with the apparent coefficient diffusion (ADC) in mm²/s. | 3 months, after surgery
For the patients who underwent surgery, evaluation of the association between size of the tumor (mm) with the apparent coefficient diffusion (ADC) in mm²/s before chimiotherapy.. | 6 months, after surgery
For the patients who underwent surgery, evaluation of the association between size of the tumor (mm) and the apparent coefficient diffusion (ADC) in mm²/s after chimiotherapy.. | 6 months, after surgery
Overall survival in years | At the end of the follow-up period (maximum 24 months).
  Time interval between the inclusion date and the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France, France

IPD SHARING:
Plan to Share IPD: No